CLINICAL TRIAL: NCT02608424
Title: Effects of Feet Mechanical Stimulation on the Inflammatory State and Cardiovascular Autonomic Profile in Patients With Parkinson's Disease
Brief Title: Effects of Feet Mechanical Stimulation on Cardiovascular Autonomic Profile and Inflammation in Parkinson's Disease
Acronym: parkgo-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: parkgo-1-ICH
Record Dates: First submitted 2015-10-27; First posted 2015-11-18 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease; Autonomic Neuropathy; Inflammation; Hypertension
Keywords: Foot mechanical stimulation; Autonomic nervous system; Inflammation; Parkinson's disease; Spectral analysis; Heart rate variability; Blood pressure variability
MeSH Terms: conditions — Parkinson Disease; Inflammation; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Foot Mechanical Stimulation (Experimental): Intervention: Foot Mechanical Stimulation (FMS) will be performed on enrolled patients every 72 hours (total 5 stimulation sessions) by a pressure-controlled mechanical stimulator (Gondola®, European Community (CE) marking n° 0476) .
  The sites of the stimulation will be the tip of the hallux and the lower big toe first metatarsal joint plantar surface. The FMS procedure consists in the application of the patient's calibrated pressure for 6 seconds, over the selected sites. Each of the 2 cutaneous sites of both feet will be mechanically stimulated. The procedure will be automatically repeated for 4 times in every subject so that the overall time of stimulation will be approximately 2 minutes.
  Interventions: Device: Foot Mechanical Stimulation (Gondola®, CE marking n° 0476)

INTERVENTIONS:
Device: Foot Mechanical Stimulation (Gondola®, CE marking n° 0476) — The feet mechanical stimulation will be performed by Gondola (Gondola®, CE marking n° 0476).
  Other Names: Pressure-controlled mechanical stimulator (Gondola®)

SUMMARY:
In the present study, investigators test the hypothesis that a controlled mechanical pressure applied on specific sites of both fore-feet (ES) can reduce the inflammatory state and arterial blood pressure in patients with Parkinson's Disease by increasing the overall parasympathetic activity and reducing vascular sympathetic modulation.

DETAILED DESCRIPTION:
Neuroinflammation may contribute to the cascade of events leading to neuronal loss in Parkinson's disease (PD) thus facilitating motor and autonomic impairment. A link between autonomic function and chronic and acute inflammation has been previously described. Specifically, active inflammatory state was associated with an overall increased sympathetic tone, whereas the parasympathetic cholinergic activation seemed to promote a decrease of inflammatory compounds in inflamed tissues. In addition, a functional link between peripheral sensory afferents and autonomic control has been reported. In a recent study it was observed that in PD patients a somatosensory activation by mechanical stimulation of specific sites of the fore-foot (effective stimulus, ES), improved gait, increased cardiac vagal modulation and decreased vascular sympathetic activity at rest. This latter effect was associated with a decline in arterial blood pressure values.

The present study is aimed at:

* Addressing the magnitude of the inflammatory state in PD patients.
* Testing the hypothesis that a change in the autonomic profile of PD patients induced by ES, consistent with cardiovascular increased parasympathetic and decreased sympathetic activities, may promote an overall reduction of the PD inflammatory state.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD characterized by a moderate/important motor impairment (Hoehn&Yhar scale 2-4)
* PD will be diagnosed according to the United Kingdom (UK) Parkinson's Disease Society Brain Bank criteria, (or on the basis of clinical criteria, Dopamine Transporter (DAT)- scan and/or MRI).

Exclusion Criteria:

* Dysautonomias and other neurodegenerative diseases
* History/familiarity with seizures
* Atrial fibrillation and other relevant cardiac rhythm disturbances
* Chronic inflammatory diseases and chronic use on anti-inflammatory drugs
* Diabetes
* Other neurological or psychiatric diseases
* Pacemakers or other electronic implants inserted into the body
* Coronary disorders, elevated intracranial blood pressure
* Assumption of drugs facilitating seizures, psychiatric drugs, alcohol abuse

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changes of Pentraxin 3 (PTX3) plasma levels induced by feet mechanical stimulation. | Blood samples will be collected at Baseline, and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  PTX3 as an index of systemic inflammatory profile will be assessed by a developed and optimized ELISA and expressed by ng/ml.
Changes of Interleukine-6 (IL-6), plasma levels induced by feet mechanical stimulation. | Blood samples will be collected at Baseline, and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  IL-6 will be tested by commercially available ELISA and immunoturbidimetric assays and expressed by ng/ml.
Changes of Tumor Necrosis Factor (TNF) plasma levels induced by feet mechanical stimulation. | Blood samples will be collected at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  TNF will be tested by commercially available ELISA and immunoturbidimetric assays and expressed by ng/ml.
Changes of C Reactive Protein (CRP) plasma levels induced by feet mechanical stimulation. | Blood samples will be collected at Baseline, and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  CRP will be tested by commercially available ELISA and immunoturbidimetric assays and expressed by mg/dl.
Changes of Heart Rate (HR) values in supine position induced by feet mechanical stimulation. | HR will be assessed in beats/min at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  Mean value of 15 minute-ECG continuous recording in supine position will be used.
Changes of Blood Pressure (BP) values in supine position induced by feet mechanical stimulation. | BP will be assessed in mmHg at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  Mean value of 5 measures obtained every 3 minutes by an Automatic-cycling non-invasive blood pressure monitor in supine position will be used.
Changes of the index of cardiac vagal modulation (HFRR, High Frequency oscillatory component of R-R interval (RR) variability at ~0.25Hz) in supine position induced by feet mechanical stimulation. | HFRR will be assessed in msec2 at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  HFRR will be obtained by the spectral analysis of R-R interval spontaneous variability in supine position.
Changes of the index of cardiac sympathetic modulation (LFRR, Low Frequency oscillatory component of R-R interval variability at ~0.10 Hz) in supine position induced by feet mechanical stimulation. | LFRR will be assessed in msec2 at baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  LFRR will be obtained by the spectral analysis of R-R interval spontaneous variability in supine position.
Changes of the index of cardiac sympatho-vagal modulation (LF/HF)RR in supine position induced by feet mechanical stimulation. | LF/HF (unit-less value) will be assessed at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  LF/HF is the ratio between LFRR index of cardiac sympathetic modulation and HFRR index of the cardiac vagal modulation obtained by the spectral analysis of R-R interval spontaneous variability.
Changes of the index of sympathetic modulation to the vessels (LFSAP) in supine position induced by by feet mechanical stimulation. | LFSAP will be assessed in mmHg2 at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  LFSAP will be quantified by spectral analysis of systolic arterial pressure variability obtained by beat by beat blood pressure non-invasive continuous recording in supine position.
Changes of plasma Norepinephrine (NE) in supine position induced by feet mechanical stimulation. | Plasma NE will be assessed in ng/L at baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  Plasma NE will be quantified by High Performance Liquid Chromatography (HPLC) with electrochemical detection (ED) from blood samples collected in supine position
Changes of plasma Epinephrine (E) in supine position induced by feet mechanical stimulation. | Plasma E will be quantified in ng/L at baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  Plasma E will be quantified by High Performance Liquid Chromatography (HPLC) and electrochemical detection (ED) from blood samples collected in supine position
Changes of Heart Rate (HR beats/min) values during 75°head-up tilt induced by feet mechanical stimulation. | HR will be assessed in beats/min at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  The mean value of 15 minute-ECG continuous recording during 75°head-up tilt will be used.
Changes of Blood Pressure (BP) values during 75°head-up tilt induced by feet mechanical stimulation. | BP will be assessed in mmHg at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  The mean value of 5 measures obtained every 3 minutes by an automatic-cycling non-invasive blood pressure monitor during 75°head-up tilt will be used.
Changes of the index of cardiac vagal modulation (HFRR, High Frequency oscillatory component of R-R interval variability at ~0.25Hz) during 75°head-up tilt induced by feet mechanical stimulation. | HFRR will be assessed in (msec2) at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  HFRR will be obtained by the spectral analysis of R-R interval spontaneous variability during 75°head-up tilt.
Changes of the index of cardiac sympathetic modulation (LFRR, Low Frequency oscillatory component of R-R interval variability at ~0.10 Hz) during 75° head-up tilt induced by feet mechanical stimulation. | LFRR will be assessed in msec2 at baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  LFRR will be obtained by the spectral analysis of R-R interval spontaneous variability during 75° head-up tilt.
Changes of the index of cardiac sympatho-vagal modulation (LF/HF)RR during 75°head-up tilt induced by feet mechanical stimulation. | LF/HF (unit-less value) will be assessed at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  LF/HF will be quantified as a ratio between LFRR index of cardiac sympathetic modulation and HFRR index of the cardiac vagal modulation obtained by the spectral analysis of R-R interval spontaneous variability during 75°head-up tilt.
Changes of the index of sympathetic modulation to the vessels (LFSAP , mmHg2) during 75°head-up tilt induced by feet mechanical stimulation. | LFSAP will be assessed in mmHg2 at Baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  LFSAP expressed will be quantified by spectral analysis of systolic arterial pressure variability obtained by beat by beat blood pressure non-invasive continuous recording during 75°head-up tilt.
Changes of plasma Norepinephrine (NE) during 75°head-up tilt induced by feet mechanical stimulation. | Plasma NE will be quantified in ng/L at baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  Plasma NE will be evaluated by High Performance Liquid Chromatography (HPLC) with electrochemical detection (ED) from blood samples collected after 5 minutes of 75°head-up tilt.
Changes of plasmatic Epinephrine (E) during 75°head-up tilt induced by feet mechanical stimulation. | Plasma E will be quantified in ng/L at baseline and 16 days from baseline (after 5 feet mechanical stimulation sessions).
  Plasma E will be evaluated by High Performance Liquid Chromatography (HPLC) and electrochemical detection (ED) from blood samples collected after 5 minutes lasting 75°head-up tilt.

SECONDARY OUTCOMES:
Changes in Unified Parkinson's Disease Rating Scale (UDPRS) induced by feet mechanical stimulation. | UDPRS will be done at baseline and 16 days from baseline, after 5 feet mechanical stimulation sessions
  UDPRS will be performed by neurologist
Changes in Timed Up and Go induced by feet mechanical stimulation. | Timed Up and Go will be evaluated at Baseline, 72 hours and 16 days from baseline after 5 feet stimulation sessions
  Timed Up and Go test will be performed before and after the feet mechanical stimulations at baseline,72 hours and 16 days from baseline (i.e. after 5 stimulations)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaello Furlan, MD, Study Director — Humanitas Research Hospital, University of Milan; Raffaello Furlan, MD, Study Chair — Humanitas Rsearch Hospital, University of Milan; Franca Barbic, MD, Principal Investigator — Humanitas Research Hospital; Humanitas University, Rozzano (MI)
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy

REFERENCES:
- [Background] Barbic F, Perego F, Canesi M, Gianni M, Biagiotti S, Costantino G, Pezzoli G, Porta A, Malliani A, Furlan R. Early abnormalities of vascular and cardiac autonomic control in Parkinson's disease without orthostatic hypotension. Hypertension. 2007 Jan;49(1):120-6. doi: 10.1161/01.HYP.0000250939.71343.7c. Epub 2006 Nov 13. PMID 17101845
- [Background] Barbic F, Galli M, Dalla Vecchia L, Canesi M, Cimolin V, Porta A, Bari V, Cerri G, Dipaola F, Bassani T, Cozzolino D, Pezzoli G, Furlan R. Effects of mechanical stimulation of the feet on gait and cardiovascular autonomic control in Parkinson's disease. J Appl Physiol (1985). 2014 Mar 1;116(5):495-503. doi: 10.1152/japplphysiol.01160.2013. Epub 2014 Jan 16. PMID 24436294
- [Background] Lee HW, Choi J, Suk K. Increases of pentraxin 3 plasma levels in patients with Parkinson's disease. Mov Disord. 2011 Nov;26(13):2364-70. doi: 10.1002/mds.23871. Epub 2011 Sep 23. PMID 21953577
- [Background] Lee JK, Tran T, Tansey MG. Neuroinflammation in Parkinson's disease. J Neuroimmune Pharmacol. 2009 Dec;4(4):419-29. doi: 10.1007/s11481-009-9176-0. Epub 2009 Oct 10. PMID 19821032
- [Background] Furlan R, Ardizzone S, Palazzolo L, Rimoldi A, Perego F, Barbic F, Bevilacqua M, Vago L, Bianchi Porro G, Malliani A. Sympathetic overactivity in active ulcerative colitis: effects of clonidine. Am J Physiol Regul Integr Comp Physiol. 2006 Jan;290(1):R224-32. doi: 10.1152/ajpregu.00442.2005. Epub 2005 Aug 25. PMID 16123227
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541
- [Background] Gademan MG, Sun Y, Han L, Valk VJ, Schalij MJ, van Exel HJ, Lucas CM, Maan AC, Verwey HF, van de Vooren H, Pinna GD, Maestri R, La Rovere MT, van der Wall EE, Swenne CA. Rehabilitation: Periodic somatosensory stimulation increases arterial baroreflex sensitivity in chronic heart failure patients. Int J Cardiol. 2011 Oct 20;152(2):237-41. doi: 10.1016/j.ijcard.2010.07.022. Epub 2010 Aug 9. PMID 20691484
- [Background] de Lau LM, Breteler MM. Epidemiology of Parkinson's disease. Lancet Neurol. 2006 Jun;5(6):525-35. doi: 10.1016/S1474-4422(06)70471-9. PMID 16713924
- [Background] Emre M. Dementia associated with Parkinson's disease. Lancet Neurol. 2003 Apr;2(4):229-37. doi: 10.1016/s1474-4422(03)00351-x. PMID 12849211
- [Background] Huse DM, Schulman K, Orsini L, Castelli-Haley J, Kennedy S, Lenhart G. Burden of illness in Parkinson's disease. Mov Disord. 2005 Nov;20(11):1449-54. doi: 10.1002/mds.20609. PMID 16007641
- [Background] Findley LJ. The economic impact of Parkinson's disease. Parkinsonism Relat Disord. 2007 Sep;13 Suppl:S8-S12. doi: 10.1016/j.parkreldis.2007.06.003. Epub 2007 Aug 16. PMID 17702630
- [Background] Allcock LM, Ullyart K, Kenny RA, Burn DJ. Frequency of orthostatic hypotension in a community based cohort of patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2004 Oct;75(10):1470-1. doi: 10.1136/jnnp.2003.029413. PMID 15377699
- [Background] Pratorius B, Kimmeskamp S, Milani TL. The sensitivity of the sole of the foot in patients with Morbus Parkinson. Neurosci Lett. 2003 Aug 7;346(3):173-6. doi: 10.1016/s0304-3940(03)00582-2. PMID 12853112
- [Background] Bernardi L, Bissa M, DeBarbieri G, Bharadwaj A, Nicotra A. Arterial baroreflex modulation influences postural sway. Clin Auton Res. 2011 Jun;21(3):151-60. doi: 10.1007/s10286-010-0099-x. Epub 2010 Dec 24. PMID 21184247
- [Background] Schmidt C, Berg D; Herting; Prieur S, Junghanns S, Schweitzer K, Globas C, Schols L, Reichmann H, Ziemssen T. Loss of nocturnal blood pressure fall in various extrapyramidal syndromes. Mov Disord. 2009 Oct 30;24(14):2136-42. doi: 10.1002/mds.22767. PMID 19768815
- [Background] Sharabi Y, Goldstein DS. Mechanisms of orthostatic hypotension and supine hypertension in Parkinson disease. J Neurol Sci. 2011 Nov 15;310(1-2):123-8. doi: 10.1016/j.jns.2011.06.047. Epub 2011 Jul 16. PMID 21762927
- [Background] Garlanda C, Bottazzi B, Bastone A, Mantovani A. Pentraxins at the crossroads between innate immunity, inflammation, matrix deposition, and female fertility. Annu Rev Immunol. 2005;23:337-66. doi: 10.1146/annurev.immunol.23.021704.115756. PMID 15771574
- [Background] Bottazzi B, Doni A, Garlanda C, Mantovani A. An integrated view of humoral innate immunity: pentraxins as a paradigm. Annu Rev Immunol. 2010;28:157-83. doi: 10.1146/annurev-immunol-030409-101305. PMID 19968561
- [Background] Mantovani A, Garlanda C, Doni A, Bottazzi B. Pentraxins in innate immunity: from C-reactive protein to the long pentraxin PTX3. J Clin Immunol. 2008 Jan;28(1):1-13. doi: 10.1007/s10875-007-9126-7. Epub 2007 Sep 9. PMID 17828584
- [Background] Furlan R, Porta A, Costa F, Tank J, Baker L, Schiavi R, Robertson D, Malliani A, Mosqueda-Garcia R. Oscillatory patterns in sympathetic neural discharge and cardiovascular variables during orthostatic stimulus. Circulation. 2000 Feb 29;101(8):886-92. doi: 10.1161/01.cir.101.8.886. PMID 10694528
- [Background] Porta A, Castiglioni P, Di Rienzo M, Bari V, Bassani T, Marchi A, Takahashi AC, Tobaldini E, Montano N, Catai AM, Barbic F, Furlan R, Cividjian A, Quintin L. Short-term complexity indexes of heart period and systolic arterial pressure variabilities provide complementary information. J Appl Physiol (1985). 2012 Dec 15;113(12):1810-20. doi: 10.1152/japplphysiol.00755.2012. Epub 2012 Oct 25. PMID 23104699